CLINICAL TRIAL: NCT06739759
Title: Prophylaxis Against Ovarian Hyperstimulation Syndrome in PCOS Women
Brief Title: Ovarian Hyperstimulation Syndrome Prevention
Acronym: OHSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, National Research centre, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ovarian hyperstimulation
Record Dates: First submitted 2024-10-23; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Hyper Stimulation Syndrome (OHSS)
Keywords: OHSS; mild; Moderate; Severe
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- antagonist (Active Comparator): patients with PCOS undergoing ICSI receiving antagonist protocol
  Interventions: Drug: Antagonist protocol for IVF
- Modified agonist with additives (Active Comparator): Patients with PCOS undergoing ICSI receiving modified agonist protocol with additives
  Interventions: Drug: Modified Agonist protocol for IVF with additive treatments as HCQ

INTERVENTIONS:
Drug: Antagonist protocol for IVF — antagonist protocol with triggering by Decapeptyl
  Other Names: Antagonist
  Arms: antagonist
Drug: Modified Agonist protocol for IVF with additive treatments as HCQ — giving additive drugs to agonist protocolas HCQ
  Other Names: modified agonist with additives
  Arms: Modified agonist with additives

SUMMARY:
Ovarian hyperstimulation is a very hazardous complication of ICSI

DETAILED DESCRIPTION:
Ovarian hyperstimulation could be mild , moderate , severe or marked

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS coming for ICSI

Exclusion Criteria:

* Women who donnot have PCOS

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with PCOS coming for ICSI
Enrollment: 300 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
prevention of OHSS | within 3 weeks
  prevention of symptoms of ovarian hyperstimulation syndrome as amount of ascites in litres by US

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, MD, Study Chair — Aljazeera Hospital
Locations (2):
- Egypt (2):
  - Aljazeerah hospital, Giza
  - Algazeerah, Giza

IPD SHARING:
Plan to Share IPD: No